CLINICAL TRIAL: NCT03606603
Title: Nutrition Insights Day Asia to Assess Hospital Malnutrition and the Routine Use of Enteral and Parenteral Nutrition in Patients Following Major Gastrointestinal Surgery
Brief Title: Nutrition Insights Day Asia
Status: Completed | Type: Observational
Sponsor: Fresenius Kabi (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: NScr-002-CNI
Record Dates: First submitted 2018-07-23; First posted 2018-07-31 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Nutritional Status; Malnutrition; Caloric Deficit; Protein Deficiency
Keywords: nutritional status; malnutrition; energy intake; protein intake; ICU; surgical ward; hospital; enteral nutrition; parenteral nutrition; nutrition
MeSH Terms: conditions — Malnutrition; Protein Deficiency; Hyperphagia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical patients: Adult patients after elective major abdominal gastrointestinal surgery with pre-existing malnutrition or who are at significant risk for malnutrition or nutrition-related complications, with indications for nutritional support

SUMMARY:
This is an observational, cross-sectional study to be conducted on the Nutrition Insights Day (NID), with retrospective review of patient medical charts. No prospective follow-up period is considered.

This study aims to obtain a contemporary overview of the nutritional status, the use of EN and/or PN and the provision of calories and proteins in patients after major elective gastrointestinal surgery with existing malnutrition or at risk of hospital malnutrition in selected Asian countries.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients after elective major abdominal gastrointestinal surgery [i.e. elective major GI resections, partial or total, especially for cancer, including: esophagectomy, gastrectomy, enterectomy (small bowel resection), colectomy, hepatectomy, pancreatectomy, resections for gall bladder or bile duct cancer (cholangiocarcinoma)] with pre-existing malnutrition or who are at significant risk for malnutrition or nutrition-related complications*, with indications for nutritional support
2. Hospitalization on SICU or major surgical ward on the NID
3. Use of EN (nutritional intake provided via tube feeding) and/or PN for at least one day before the NID
4. If patient received oral nutrition (ON) or oral nutrition supplements (ONS) during the observational phase from day -5 to day -2, complete and reliable data of daily caloric and protein intake is available
5. Latest surgical intervention ≤ 10 days before NID

Exclusion Criteria:

1. Patients with burn injuries
2. Patients requiring postsurgical mechanical ventilation and sedation on the NID
3. Patients receiving ON and/or ONS at any quantity on the day before the NID
4. Patients requiring emergency procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients after elective major abdominal gastrointestinal surgery with pre-existing malnutrition or who are at significant risk for malnutrition or nutrition-related complications, with indications for nutritional support
Sampling Method: Non-Probability Sample
Enrollment: 590 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Proportion of surgical patients with a caloric / protein deficit receiving EN and/or PN on the day before the NID in selected Asian countries. | On the day before the Nutrition Insights Day (day -1)
  Caloric / protein deficit, i.e., difference between energy / protein target per day and actually administered energy/protein

SECONDARY OUTCOMES:
Absolute and relative caloric and protein balance | On the day before the Nutrition Insights Day (day -1)
  Absolute and relative caloric and protein balance
Distribution within subcategories of caloric / protein balance | On the day before the Nutrition Insights Day (day -1)
  Distribution within subcategories of caloric / protein balance
Cumulative (absolute/ relative) caloric and protein balance | On the day before the Nutrition Insights Day (day -1)
  Cumulative (absolute/ relative) caloric and protein balance
Categorical, absolute and relative caloric balance based on standardized target intake (sensitivity analysis) | On the day before the Nutrition Insights Day (day -1)
  Categorical, absolute and relative caloric balance based on standardized

CONTACTS AND LOCATIONS:
Overall Officials: John F Stover, M.D., Study Chair — Fresenius Kabi
Locations (89):
- India (27):
  - Manipal Hospital, Bangalore
  - Bombay Hospital, Bombay
  - Apollo Hospitals, Chennai
  - SIMS (SRM Institutes for Medical Science), Chennai
  - G. Kuppuswamy Naidu Memorial Hospital, Coimbatore
  - Max Super Speciality Hospital, Dehli
  - Sir Ganga Ram Hospital, Dehli
  - AMRI Hospital, Dhakuria
  - Fortis Memorial Research Institute, Gūrgaon
  - Medanta Medicity Hospital, Gūrgaon
  - Care Hospital, Hyderabad
  - Rukmani Birla Hospital, A Unit of CMRI, Jaipur
  - Rukmani Birla Hospital, Jaipur
  - Apollo Gleneagles Hospitals Ltd., Kolkata
  - Dayanand Medical College and Hospital, Ludhiana
  - Fortis Hospital, Mohali
  - Max Superspecialty Hospital, Mohali
  - B. Y. L. Nair Charitable Hospital & Topiwala National Medical College, Mumbai
  - S.L Raheja - A Fortis Associate Hospital, Mumbai
  - BLK Super Specialty Hospital, New Delhi
  - Jawaharlal Institute Of Post Graduate Medical Education Medical Education and Research (JIPMER), Puducherry
  - Deenanath Mangeshkar Hospital, Pune
  - Ruby Hall Clinic, Pune
  - Krishna Institute of Medical Sciences, Secunderabad
  - Surat Institute of Digestive Sciences, Sūrat
  - Geetanjali Medical College, Udaipur
  - Christian Medical College & Hospital, Vellore
- Indonesia (9):
  - Cipto Mangunkusumo Hospital, Jakarta
  - Dharmais Cancer Center, Jakarta
  - Rumah Sakit Persahabatan, Jakarta
  - Siloam Hospitals Kebon Jeruk, Jeruk
  - Kariadi Hospital, Semarang
  - Telogorejo Hospital, Semarang
  - Mitra Keluarga Waru Hospital, Waru
  - Bethesda Hospital, Yogyakarta
  - Sardjito Hospital, Yogyakarta
- Philippines (18):
  - Capitol University Medical Center, Cagayan de Oro
  - Cebu Doctors University Hospital, Cebu City
  - Perpetual Succour Hospital, Cebu City
  - De La Salle University Medical Center, Dasmariñas
  - Southern Philippines Medical Center, Davao City
  - Makati Medical Center, Makati City
  - Asian Hospital and Medical Center, Manila
  - Dr. Jose R.Reyes Memorial Medical Center, Manila
  - Manila Doctors Hospital, Manila
  - Philippine General Hospital, Manila
  - St. Luke's Medical Center Global City, Manila
  - University of Santo Tomas, Manila
  - The Medical City, Pasig
  - East Avenue Medical Center, Quezon City
  - National Kidney and Transplant Institute, Quezon City
  - Quirino Memorial Medical Center, Quezon City
  - St. Luke's Medical Center, Quezon City
  - Jose B.Lingad Memorial Regional Memorial Hspl, San Fernando City
- South Korea (9):
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Hospital, Daegu
  - National Cancer Center, Goyang-si
  - Chungnam National University Hospital, Jungnam
  - Seoul National University Bundang Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Sungkunkwan University Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Ulsan University Hospital, Asan Medical Center, Ulsan
- Taiwan (9):
  - Changhua Christian Medical Foundation Changhua Christian Hospital, Chang-hua
  - Chang Gung Memorial Hospital- Kaoshiung Branch, Kaohsiung City
  - E-DA Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital, Linkou District
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Thailand (10):
  - Bhumibol Adulyadej Hospital, Bangkok
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Rajavithi Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Srinakarin Hospital, Bangkok
  - Thammasat University Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Songkla Nakarin Hospital, Hat Yai
  - Siriraj Hospital, Phuket
  - Surin Hospital, Surin
- Vietnam (7):
  - 108 Military Central Hospital, Hanoi
  - Bach Mai Hospital, Hanoi
  - Cho Ray Hospital, Ho Chi Minh City
  - HCM city University Medical Center, Ho Chi Minh City
  - People's Hospital 115, Ho Chi Minh City
  - Thong Nhat Hospital, Ho Chi Minh City
  - Hue Central Hospital, Huế

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Detsky AS, McLaughlin JR, Baker JP, Johnston N, Whittaker S, Mendelson RA, Jeejeebhoy KN. What is subjective global assessment of nutritional status? JPEN J Parenter Enteral Nutr. 1987 Jan-Feb;11(1):8-13. doi: 10.1177/014860718701100108. PMID 3820522
- [Result] Higashiguchi T, Arai H, Claytor LH, Kuzuya M, Kotani J, Lee SD, Michel JP, Nogami T, Peng N. Taking action against malnutrition in Asian healthcare settings: an initiative of a Northeast Asia Study Group. Asia Pac J Clin Nutr. 2017 Mar;26(2):202-211. doi: 10.6133/apjcn.022016.04. PMID 28244696
- [Result] Ho JW, Wu AH, Lee MW, Lau SY, Lam PS, Lau WS, Kwok SS, Kwan RY, Lam CF, Tam CK, Lee SO. Malnutrition risk predicts surgical outcomes in patients undergoing gastrointestinal operations: Results of a prospective study. Clin Nutr. 2015 Aug;34(4):679-84. doi: 10.1016/j.clnu.2014.07.012. Epub 2014 Aug 1. PMID 25175758
- [Result] Jia ZY, Yang J, Tong DN, Peng JY, Zhang ZW, Liu WJ, Xia Y, Qin HL. Screening of nutritional risk and nutritional support in general surgery patients: a survey from Shanghai, China. Int Surg. 2015 May;100(5):841-8. doi: 10.9738/INTSURG-D-14-00245.1. PMID 26011204
- [Result] Kondrup J, Rasmussen HH, Hamberg O, Stanga Z; Ad Hoc ESPEN Working Group. Nutritional risk screening (NRS 2002): a new method based on an analysis of controlled clinical trials. Clin Nutr. 2003 Jun;22(3):321-36. doi: 10.1016/s0261-5614(02)00214-5. PMID 12765673
- [Result] Linthicum MT, Thornton Snider J, Vaithianathan R, Wu Y, LaVallee C, Lakdawalla DN, Benner JE, Philipson TJ. Economic burden of disease-associated malnutrition in China. Asia Pac J Public Health. 2015 May;27(4):407-17. doi: 10.1177/1010539514552702. Epub 2014 Oct 8. PMID 25301845
- [Result] Liu X, Xu P, Qiu H, Xu D, Li W, Zhan Y, Li Y, Chen Y, Zhou Z, Sun X. Preoperative Nutritional Deficiency Is a Useful Predictor of Postoperative Outcome in Patients Undergoing Curative Resection for Gastric Cancer. Transl Oncol. 2016 Dec;9(6):482-488. doi: 10.1016/j.tranon.2016.09.008. Epub 2016 Oct 24. PMID 27788388
- [Result] Nakahara S, Nguyen DH, Bui AT, Sugiyama M, Ichikawa M, Sakamoto T, Nakamura T. Perioperative nutrition management as an important component of surgical capacity in low- and middle-income countries. Trop Med Int Health. 2017 Jul;22(7):784-796. doi: 10.1111/tmi.12892. Epub 2017 Jun 13. PMID 28510990
- [Result] Norman K, Pichard C, Lochs H, Pirlich M. Prognostic impact of disease-related malnutrition. Clin Nutr. 2008 Feb;27(1):5-15. doi: 10.1016/j.clnu.2007.10.007. Epub 2007 Dec 3. PMID 18061312
- [Result] Sun Z, Kong XJ, Jing X, Deng RJ, Tian ZB. Nutritional Risk Screening 2002 as a Predictor of Postoperative Outcomes in Patients Undergoing Abdominal Surgery: A Systematic Review and Meta-Analysis of Prospective Cohort Studies. PLoS One. 2015 Jul 14;10(7):e0132857. doi: 10.1371/journal.pone.0132857. eCollection 2015. PMID 26172830
- [Result] Vallejo KP, Martinez CM, Matos Adames AA, Fuchs-Tarlovsky V, Nogales GCC, Paz RER, Perman MI, Correia MITD, Waitzberg DL. Current clinical nutrition practices in critically ill patients in Latin America: a multinational observational study. Crit Care. 2017 Aug 25;21(1):227. doi: 10.1186/s13054-017-1805-z. PMID 28841885
- [Result] Waitzberg DL, Caiaffa WT, Correia MI. Hospital malnutrition: the Brazilian national survey (IBRANUTRI): a study of 4000 patients. Nutrition. 2001 Jul-Aug;17(7-8):573-80. doi: 10.1016/s0899-9007(01)00573-1. PMID 11448575
- [Result] Zhong JX, Kang K, Shu XL. Effect of nutritional support on clinical outcomes in perioperative malnourished patients: a meta-analysis. Asia Pac J Clin Nutr. 2015;24(3):367-78. doi: 10.6133/apjcn.2015.24.3.20. PMID 26420176